CLINICAL TRIAL: NCT05507983
Title: Tranexamic Acid During Excisional Burn Surgery
Acronym: TRANEX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Collaborators: Association of Dutch Burn Centres (Other); Martini Hospital Groningen (Other); Red Cross Hospital Beverwijk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL69319.100.20; WO 19.102 (Other Grant/Funding Number: Dutch Burn Foundation)
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Burns; Blood Loss, Surgical; Blood Loss; Tranexamic Acid; Burn Excisional Surgery
Keywords: Blood loss; Tranexamic Acid; Burn excisional surgery; Burns
MeSH Terms: conditions — Burns; Blood Loss, Surgical; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid arm (Experimental): Tranexamic acid 1500 mg dissolved in 100 ml sodium chloride, once, directly after anesthetizing the participant.
  In participants with renal insufficiency (creatinine >120 umol/L) the dose will be reduced to 1000 mg.
  Interventions: Drug: Tranexamic acid
- Placebo arm (Placebo Comparator): 100ml sodium chloride 0.9%, once, directly after anesthetizing the participant.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic acid 1500 mg
  Arms: Tranexamic acid arm
Drug: Placebo — Placebo, sodium chloride 0.9%
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to access the efficacy of the drug tranexamic acid in reducing blood loss during burn excision surgery.

DETAILED DESCRIPTION:
This study is a double-blinded, randomized placebo-controlled trial. After informed consent patients will be randomized in either the placebo or the tranexamic acid group (1500 mg). The intervention will be conducted during burn excisional surgery. First, the participant with be anesthetized, whereafter the study medication is administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for burn excisional surgery
* An expected blood loss of ≥250ml based on the estimation by the performing surgeon on the basis of: (1) ≥ 2 % body surface area excision planned (100-200 cc / % total body surface area, (2) operation technique used (some techniques show more blood loss than others), (3) time after burn trauma (i.e. expected healing)
* ≥18 year
* informed consent of patient or legal representative
* Patients or legal representative should have enough knowledge of Dutch to provide informed consent

Exclusion Criteria:

* Patients with a recorded coagulopathy in their history
* The use of anticoagulants (except acetylsalicylic acid or (intensive) prophylaxis low molecular weight heparin >12 hours before surgery)
* Severe kidney failure (creatinine >500 μmol/L)
* Allergy for tranexamic acid
* Diagnosis of acute venous-/arterial thrombosis within 3 months before inclusion
* Diffuse intravascular coagulation (based on the diffuse intranasal coagulation-score >5)
* Pregnancy
* Active breastfeeding
* History of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Blood loss | During burn excisional surgery
  Volume of blood loss measured during surgery.

SECONDARY OUTCOMES:
Hospital Mortality | During total admittance of the patient
  % of mortality in patients participating in this study.
Length of stay in days | The length of stay will be evaluated after 3 months after inclusion. If, after 3 months, the patient is still admitted, the status of hospitalisation will be check after an addition 3 months.
  Number of days admitted after burn trauma.
Graft failure in % of total graft | During burn excisional surgery
  % of graft failure of the total graft.
Cardiopulmonary complications | Within the first 30 days after burn excisional surgery
  i.e. pulmonary embolism, arterial embolism.
Neurologic complications | Within the first 30 days after burn excisional surgery
  i.e. stroke of epilepsy
The need for escape medication | During burn excisional surgery
  Out of protocol administration of tranexamic acid based on massive blood loss.
Extend of fibrinolysis during burn excisional surgery | During burn excisional surgery
  Measured by ROTEM analysis
Strength of blood clot | During burn excisional surgery
  Analysis will be performed using (electron) microscope to investigate: strength, thickness, structure of fibrin, fibrin clot networks and cell disposition within the blood clot.
Transfusion requirements | Perioperative, within the first day after surgery.
  Number of transfusions in the perioperative phase.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Red Cross Hospital, Beverwijk, North Holland
  - Maasstad Hospital, Rotterdam, South Holland
  - Martini Hospital, Groningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gigengack RK, Slob J, Vries AM, Bosma E, Loer SA, Koopman JSHA, van der Vlies CH. Efficacy of tranexamic acid versus placebo in reducing blood loss during burn excisional surgery: a multi-center, double-blind, parallel, randomized placebo-controlled clinical trial (TRANEX). Trials. 2024 Aug 2;25(1):520. doi: 10.1186/s13063-024-08332-1. PMID 39095919